CLINICAL TRIAL: NCT02758782
Title: COmparison of the Effect of Treatment With NSAIDs Added to Anti-TNF Therapy Versus Anti-TNF Therapy Alone on Progression of StrUctural Damage in the Spine Over Two Years in Patients With ankyLosing Spondylitis: a Randomized Controlled Multicentre Trial
Brief Title: NSAIDs Added to Anti-TNF Therapy Versus Anti-TNF Therapy Alone on Progression of Structural Damage in Ankylosing Spondylitis
Acronym: CONSUL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Denis Poddubnyy, Prof Dr Denis Poddubnyy, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONSUL2016
Record Dates: First submitted 2016-04-20; First posted 2016-05-02 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — golimumab; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Golimumab monotherapy (Active Comparator): Treatment with 50 mg Golimumab subcutaneous once monthly
  Interventions: Biological: Golimumab
- Golimumab combined with Celecoxib (Active Comparator): Treatment with Golimumab 50 mg subcutaneous once monthly in combination with Celecoxib 400 mg orally every day
  Interventions: Biological: Golimumab; Drug: Celecoxib

INTERVENTIONS:
Biological: Golimumab
  Other Names: Simponi
Drug: Celecoxib
  Other Names: Celebrex
  Arms: Golimumab combined with Celecoxib

SUMMARY:
To evaluate the impact of treatment with a non-steroidal anti-inflammatory drug (NSAID) - Celecoxib - when added to anti-tumour necrosis factor (TNF) therapy - Golimumab - as compared to anti-TNF therapy (Golimumab) alone on progression of structural damage in the spine over two years in patients with ankylosing spondylitis (AS).

DETAILED DESCRIPTION:
The aim of the proposed trial is to evaluate the efficacy of combined treatment with a non-steroidal anti-inflammatory drug (NSAID) added to anti-tumour necrosis factor (TNF) therapy as compared to anti-TNF therapy alone on progression of structural damage in the spine over two years in patients with ankylosing spondylitis (AS). The trial consists of two phases. In the phase I (run-in phase), patients with active AS despite treatment with NSAIDs and elevated C-reactive protein will be included and treated with a TNF blocker (golimumab). Patients with good clinical response to golimumab at week 12 will be eligible for the phase II (core phase) of the study and will be randomized 1:1 to 1) golimumab + celecoxib (experimental intervention) for 2 years (weeks 12-108) or 2) golimumab alone (control intervention) also for 2 years. The primary outcome parameter will be the absolute progression of the modified Stoke Ankylosing Spondylitis Spine Score (mSASSS) - currently a standard of structural spinal damage progression evaluation in AS - over two years of therapy (weeks 12-108).

ELIGIBILITY:
Major Inclusion Criteria:

* Definite diagnosis of AS according to the "modified New York criteria".
* History of an inadequate response to ≥2 NSAIDs taken for at least 2 weeks each.
* Active disease as defined by a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) value of ≥4 at screening.
* Presence of at least one of the following risk factors for radiographic spinal progression:

  1. Elevated C reactive protein (CRP; >5mg/l) at screening at the absence of reasons for elevated CRP other than AS;
  2. Presence of ≥ 1 syndesmophyte on prior X-rays of the spine.
* Subject is a candidate for anti-TNF therapy based on the Investigator's opinion.
* Subject is able and willing to give a written informed consent and comply with the requirements of the study protocol. Only patients who give written informed consent will be included in the trial.
* If female: either unable to bear children (postmenopausal for at least 1 year or surgically sterile) or is willing and able to practice a reliable method of contraception throughout the study and 6 months after

Inclusion Criterion for Phase II (randomized part of the study):

- adequate response to Golimumab during Phase I (referred to as decline in BASDAI)

Major Exclusion Criteria:

* For female subjects: pregnancy or lactating
* subjects with chronic inflammatory articular disease other than spondyloarthritis / AS or systemic autoimmune disease, e.g. systemic lupus erythematosus, Sjögren´s syndrome, rheumatoid arthritis.
* history of inadequate response to anti-TNF-therapy
* intolerability/hypersensitivity to one of the drugs or other components of the study medication
* presence ot total spinal ankylosis
* contraindications to anti-TNF-therapy (current or remitting clinical significant infections, tuberculosis, viral hepatitis, HIV; malignancies; demyelinating disease; vaccination with live vaccine within 3 months before, during and until 6 months after study)
* (relative) contraindications to Celecoxib therapy (uncontrolled arterial hypertension, high cardiovascular risk / history of cardiovascular events; history of gastrointestinal ulcers or relevant bleeding; known M. Crohn or ulcerative colitis)
* diagnosis of fibromyalgia
* significant lab abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2016-09; Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Absolute progression of the modified Stoke Ankylosing Spondylitis Spine Score (mSASSS) over two years of therapy (weeks 12-108) in the Phase II (core phase) of the trial | 2 years
  Absolute progression of the modified Stoke Ankylosing Spondylitis Spine Score (mSASSS) over two years of therapy (weeks 12-108) in the Phase II (core phase) of the trial

SECONDARY OUTCOMES:
New syndesmophyte formation or progression of existing syndesmophytes | 2 years
  New syndesmophyte formation or progression of existing syndesmophytes
Improvement of disease activity (BASDAI) | 2 years
  Improvement of disease activity (BASDAI)
Improvement of disease activity (ASDAS) | 2 years
  Improvement of disease activity (ASDAS)
Improvement of function (BASFI) | 2 years
  Improvement of function (BASFI)
Improvement of axial mobility (BASMI) | 2 years
  Improvement of axial mobility (BASMI)
Improvement of quality of life measures (ASAS Health Index) | 2 years
  Improvement of quality of life measures (ASAS Health Index)
Change of the enteric microbiome profile at week 108 in comparison to baseline | 2 years
  Change of the enteric microbiome profile at week 108 in comparison to baseline
Change of Berlin MRI score (SUBSTUDY) | 2 years
  Change of Berlin MRI score (SUBSTUDY)
Adverse events (AE), serious AE and AE of interest until end of study | 2 years
  Adverse events (AE), serious AE and AE of interest until end of study

CONTACTS AND LOCATIONS:
Overall Officials: Denis Poddubnyy, Prof. Dr., Principal Investigator — Head of Dpt. for Rheumatology at Charite, Campus Benjamin Franklin
Locations (19):
- Germany (19):
  - Rheumapraxis Kupka, Altenburg
  - Rheumapraxis Bayreuth Dr. Ochs, Bayreuth
  - Charite Universitaetsmedizin - Dpt. Rheumatology at Campus Charite Mitte, Berlin
  - Rheumatologische Schwerpunktpraxis, Berlin
  - Rheumatologische Praxis Dr. Karberg/Brandt, Berlin
  - Charite Universitaetsmedizin, Dpt. of Rheumatology at Campus Benjamin Franklin, Berlin
  - MVZ Drs. Mielke, Berlin
  - Rheumapraxis Dr. Zinke, Berlin
  - Schlossparkklinik, Dpt. of Rheumatologie, Berlin
  - Rheumatologische Schwerpunktpraxis an den Kreiskliniken, Burghausen
  - Universitätsklinikum Köln, Rheumatologie, Cologne
  - Centrum für innovative Diagnostik und Therapie Rheumatologie/Immunologie (CIRI), Frankfurt am Main
  - Praxis Dr Kühne, Haldensleben I
  - Medizinische Hochschule, Rheumatologie, Hanover
  - Rheumazentrum Ruhrgebiet, Herne
  - Rheumapraxis Magdeburg, Magdeburg
  - Klinikum Rechts der ISAR (TU München), München
  - Rheumapraxis Dr. Jacki, Tübingen
  - University of Tuebingen, Dpt. Rheumatology, Tübingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Proft F, Muche B, Listing J, Rios-Rodriguez V, Sieper J, Poddubnyy D. Study protocol: COmparison of the effect of treatment with Nonsteroidal anti-inflammatory drugs added to anti-tumour necrosis factor a therapy versus anti-tumour necrosis factor a therapy alone on progression of StrUctural damage in the spine over two years in patients with ankyLosing spondylitis (CONSUL) - an open-label randomized controlled multicenter trial. BMJ Open. 2017 Jun 10;7(6):e014591. doi: 10.1136/bmjopen-2016-014591. PMID 28601821